CLINICAL TRIAL: NCT07325058
Title: Exploration of the Effect, and Their Duration, of Different Frequency Transcutaneous Auricular Vagal Nerve Stimulation on Sensory Perception.
Brief Title: Tonic Pain and Transauricular Vagal Nerve Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Laura De Herde, Principle Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: N-20230022-5
Record Dates: First submitted 2025-12-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Experimental Pain in Healthy Human Subjects
Keywords: cross-over; taVNS

STUDY DESIGN:
Intervention Model Description: Burst-taVNS, active-control (electrical stimulation of the earlobe) or sham will be administred to the participant on one of the three visits. Order of stimulation condition will be randomly selected and counter-balanced across participants (minding sex at birth).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Electrodes for the different stimulation conditions will be applied during all three visits regardless of which stimulation is active. Wiring of the electrodes is the same but labelled with 'A' or 'B'. Corresponding stimulation condition will not be known to the experimenter (that is also analyzing the data) until after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- taVNS (Experimental): Bursts of 25Hz occuring for 3.4sec every 29.4sec for 40min.
  Interventions: Device: taVNS
- Earlobe Stimulation (Active Comparator): Bursts of 25Hz occuring for 3.4sec every 29.4sec for 40min.
  Interventions: Device: Earlobe Stimulation
- Sham (Placebo Comparator): No stimulation.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: taVNS — Two-headed ball-point electrode which is placed in the concha cymba.
  Arms: taVNS
Device: Earlobe Stimulation — Circular urface adhering electrodes will be attached to either facet of the earlobe.
  Arms: Earlobe Stimulation
Device: Sham (No Treatment) — Circular surface adhesive electrodes will be placed on either facet of the earlobe. No current will pass through the electrodes.
  Arms: Sham

SUMMARY:
This study aims to explore the effect of burst-taVNS (electric stimulation of the concha cymba) on tonic (capsaicin-induced skin pain) and acute (pressure pain sensitivity) experimental pain and cardioception. Primary outcomes include pain intensity. Secondary outcomes include sensory thresholds, resting heart rate (EKG), pupillary measurements and conditioned pain modulation.

DETAILED DESCRIPTION:
Across 3 visits, each lasting around 2.5hours, burst-taVNS (electrical stimulation of the concha cymba) will be compared to active-control (electrircal stimulation of the earlobe) and sham (no current) stimulation, two gold-standard controls. Assessments of outcomes will occur before capsaicin application and before, twice during and after electrical ear stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Speak and understand English
* 18-60 years old.

Exclusion Criteria:

* Pregnant and/or breastfeeding
* Regular use of cannabis, opioids or other drugs
* Current or previous neurologic, musculoskeletal, mental, or other illnesses (e.g., brain or spinal cord injuries, degenerative neurological disorders, major depression, cardiovascular disease, chronic lung disease, etc.)
* Current regular (once or more a week) use of analgesic medication or other medication which may affect the trial (including paracetamol and NSAIDs)
* Recent history of acute pain particularly in the lower limbs
* Abnormally disrupted sleep in 24 hours preceding experiment
* Contraindications to electric stimulation application (history of epilepsy, metal implants in head or jaw, etc.)
* Lack of ability to cooperate
* Contraindications for capsaicin including an intolerance chili consumption and burns or wounds to the application site.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From when capsaicin is applied to the end of the experiment in 5 min intervals.
  Capaisin is a topically administered tonic pain model. Stemming from its chilly-origin, pain induced ressembels heat/light burning sensation which increases within 20minute of application to the forearm, before it plateaus. Associated pain can be stopped immediately by applying ice/cold water. Participants will be asked to rate (using a scale from 0 denoting no pain, to 10 denoting maximal pain) the intensity of the pain in 5 min time intervals.

SECONDARY OUTCOMES:
Pressure Pain Detection Threshold | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  Using the computerized pressure pain algometer tool (Nocitech, Aalborg, Denmark), cuffs placed on the calves of participants wll inflate at a consistent rate. Participants are instructed to rate the pain experiences using a visual analogue scale (VAS) and to press a button when the pain becomes intolerable. The VAS ranges from 0 denoting no pain, to 10 denoting maximal pain. Pain detection, namely the kPa where the VAS is at 1cm, and the pain tolerance, namely the kPa when the deflation-button is pressed, will be acquired.
Conditioned Pain Modulation Effect | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  Using the computerized pressure pain algometer tool (Nocitech, Aalborg, Denmark), cuffs placed on the calves of participants wll inflate at a consistent rate. Whilst participants have a constant pressure applied to their non-dominant leg, they are instructed to rate the pain experienced on the dominant leg as the cuff slowly inflates using a visual analogue scale (VAS) and to press a button when the pain becomes intolerable. The VAS ranges from 0 denoting no pain, to 10 denoting maximal pain. Conditioned pain detection, namely the kPa where the VAS is at 1cm, will be acquired.
Pressure Pain Perception | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  Trapezius pressure pain perception will be acquired using a handheld pressure algometer (Somedic, Solna, Sweden). Perpendicular to the musle and halfway between the acrominion and the processus spinous vertebrae, the 1cm2 probe will be applied at a constant rate. When particpants first feel pressure pain, they will respond with a button-press.
Pupillary Light Reflex | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  Using the Neurolight, per pupil, a 3s light reflex will be acquired. This refers to the reflex following the exposure to a light flash.
Electrocardiography | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  Using a 3-lead system (reference electrode on the clavicle, whilst the other two leads reside on the sternum and V4), resting state electrocardiography will be acquired.
Cardioception Accuracy | Before Capsaicin application and at 3 time intervals from when the ear stimulation (taVNS, Active Control or Sham) is applied: before, as the stimulation starts and halfway during (at min 20).
  The ability to perceive your heart beats is described as cardioception. One means by which to assess this ability is the 'heartbeat couting task'. Herein, using a queue, participants are tasked to count their heartbeats in 3 undislosed and randomized durations (25, 35 and 35s). This value is then compare to the actual number of beats during each time interval, which is acquired via electrocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Neuroplasticity and Pain, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
There is only one researcher working on this project. Information will not be shared.